CLINICAL TRIAL: NCT03842267
Title: A Multicenter, Randomized, Placebo-controlled, Parallel Group, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of Gemigliptin 50mg in Patients With Type 2 Diabetes Who Have Inadequate glycemIc Control With Dapagliflozin and Metformin (SOLUTION Study)
Brief Title: A Study to Evaluate the Efficacy and Safety of Gemigliptin in Type 2 Diabetes Who Have Inadequate GlycemIc Control With Dapagliflozin and Metformin (SOLUTION Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-DPCL019
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemigliptin 50mg (Active Comparator)
  Interventions: Drug: Gemigliptin 50mg
- Gemigliptin Placebo (Placebo Comparator)
  Interventions: Drug: Gemigliptin Placebo

INTERVENTIONS:
Drug: Gemigliptin 50mg — * The subjects should visit a study site 9 times during the treatment period for about 52 weeks in total.
  * Background therapy should be administered at the same time every day, keeping the same dosage administered before the study, according to the following criteria:
    1. Dapagliflozin 10 mg / day
    2. Metformin ≥ 1,000 mg / day
  Arms: Gemigliptin 50mg
Drug: Gemigliptin Placebo — * The subjects should visit a study site 9 times during the treatment period for about 52 weeks in total.
  * - The subjects should visit a study site 9 times during the treatment period for about 52 weeks in total.
  * Background therapy should be administered at the same time every day, keeping the same dosage administered before the study, according to the following criteria:
    1. Dapagliflozin 10 mg / day
    2. Metformin ≥ 1,000 mg / day
  Arms: Gemigliptin Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of gemigliptin 50 mg orally administered once daily for 24 weeks compared with placebo in patients with type 2 diabetes mellitus who have inadequate glycemic control with dapagliflozin and metformin

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus of upper 19 years old at the time of Visit 1 (Screening)
2. Visit 1 (Screening) Patients who had taken Dapagliflozin 10mg/day and Metformin(≥1000mg/day) more than 8 weeks and who have inadequate blood glucose control at Visit 1 (Screening)
3. Patients who have signed an informed consent themselves after receiving explanation about the objectives, methods, effects, etc. of the clinical study
4. Patients who are applicable to one of the three in the following. 1) Surgically infertile patients 2) Postmenopausal female patients of ≥45 years of age for whom ≥2 years elapsed since their last menstruation 3) Premenopausal fertile female patients or surgically non-infertile male patients who have agreed to use at least 2 kinds of contraceptive measures (certainly including one of the barrier methods) to avoid pregnancy until 14 days after the last dose of the investigational product

   * Barrier methods: Condom, Diaphragm, Cervical cap(Pessary), Spermicide
   * Hormonal methods: Pills, Injection(Depot), Skin patch, Hormonal implant(Implanon), Vaginal ring
   * Intrauterine Devices(IUDs): Cooper IUD(Loop), Hormonal IUD(Mirena)
   * Natural methods: Basic body temperature, Ovulation period, Coitus interruptus, Abstinence

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus, Diabetic ketoacidosis, Metabolic acidosis Diabetic coma, Diabetic pre-coma
2. Patients with Gestational diabetes, or secondary diabetes
3. Patients with Body Mass Index(BMI) >40 kg/m2 at the time of Visit 1(Screening)
4. Patients with a history of the following

   * Patients with NYHA Class II~IV congestive heart failure or arrhythmia requiring treatment at the time of Visit 1(Screening)
   * Patients whose TSH level is out of the normal range and who have thyroidal dysfunction requiring drug therapy at the time of Visit 1(Screening) (However, those who have been taking thyroid hormone at a fixed dose since previous 4 weeks prior to Visit 1(Screening) and whose TSH level is within the normal range can participate in the study.)
   * Patients with a glomerular filtration rate (eGFR) less than 45 mL/min /1.73 m2, moderate of severe stage renal disease, end-stage renal disease, dialysis at the time of Visit 1(Screening)
   * Patients who are receiving intravenous iodine contrast agents within 48 hours prior to Visit 1(Screening) or planned during the clinical trial period (eg, intravenous urography, venous cholangiography, angiography, computed tomography using contrast media, etc.).
   * Patients with pulmonary embolism, severe pulmonary dysfunction, or who are susceptible to be accompanied by hypoxemia at the time of Visit 1(Screening)
   * Patients on dehydration, diarrhea, and vomiting at the time of Visit 1(Screening)
   * Patients with pituitary insufficiency or adrenal insufficiency at the time of Visit 1(Screening)
   * Patients with a history of myocardial infarction, unstable angina, and Cerebrovascular disease within 12 weeks prior to Visit 1(Screening)
   * Patients who had had a surgical operation within 4 weeks prior to Visit 1(Screening) (excluding minor surgeries without restriction on food and fluid intake) or who are scheduled to have a significant surgery during the study period
   * Patients with a history of alcoholism or drug addiction within 1 years prior to Visit 1(Screening)
   * Patients with a history of malignant tumors within 5 years prior to Visit 1(Screening). However, patients with basal cell or squamous cell skin cancer, or in situ cervical cancer treated properly can participate in the study.
5. Patients with the outcomes of the laboratory tests performed at Visit 1(Screening) applicable to the criteria below

   * Bilirubin >2 × upper limit of normal(ULN)
   * AST/ALT >3 × ULN
6. Patients with a history of hypersensitivity reactions to the drugs below

   * Dipeptidyl-peptidase4(DPP4) inhibitors
   * Sodium/glucose co transport-2(SGLT-2) inhibitor
   * Biguanides
7. Patients who were administered the drugs below

   * Patients who had been administered anti-obesity drugs within 12 weeks prior to Visit 1(Screening)
   * Patients who had been administered insulin or GLP-1 analogues within 8 weeks prior to Visit 1(Screening)
   * Patients who had been being administered glucocorticoids, Strong CYP3A4 inducers continuously within 2 weeks prior to Visit 1(Screening) or who are required to take glucocorticoids continuously in the future
8. Patients with positive Serologic results of HBsAg, HCV Ab, HIV Ab test within 4 weeks prior to Visit 1 (Screening) or at Visit 1 (Screening)
9. Patients who have undergone bariatric surgery within the 1 year prior to Visit 1 (Screening) or are scheduled during the trial
10. Patients with a genetic problems such as Galactose intolerance, Lapp lactose deficiency, Glucose-galactose malabsorption)
11. Female patients who are pregnant or lactating
12. Patients who have an experience of participation in another clinical study within 12 weeks prior to Visit1(screening)
13. Patients who are otherwise considered to be ineligible for this study on investigators' judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline HbA1c at week 24 | Baseline (week 0) and week 24

CONTACTS AND LOCATIONS:
Locations (1):
- LG chem, Seoul, Gangseo-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No